CLINICAL TRIAL: NCT02899676
Title: Neural Bases of Arithmetic Processing: MRIf Study in Adults and Children
Brief Title: Cerebral Bases of Arithmetics Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013.801
Record Dates: First submitted 2016-09-02; First posted 2016-09-14 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Neural Bases of Arithmetic Processing
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy subjects aged 18 to 24 (Experimental): Subjects without neurological or psychiatric history
  Interventions: Other: neuropsychological testing; Other: functional magnetic resonance imaging; Other: simple arithmetic operations
- Healthy subjects aged 8 to 11 (Experimental): Subjects without neurological or psychiatric history
  Interventions: Other: neuropsychological testing; Other: functional magnetic resonance imaging; Other: simple arithmetic operations
- Healthy subjects aged 12 to 14 (Experimental): Subjects without neurological or psychiatric history
  Interventions: Other: neuropsychological testing; Other: functional magnetic resonance imaging; Other: simple arithmetic operations

INTERVENTIONS:
Other: neuropsychological testing
Other: functional magnetic resonance imaging
  Other Names: IRMf
Other: simple arithmetic operations

SUMMARY:
The aim of this study was to identify neural correlates involved in arthmetics processing in adults and children aged 8 to 14 with normal cognitive function. Brain area will be identified by functional magnetic resonance imaging (IRMf).

ELIGIBILITY:
Inclusion Criteria:

* children aged 8 to 14 with parents' consent
* adults aged 18 to 24
* right-handed
* affiliated to the French social security

Exclusion Criteria:

* known neurological disorders including epilepsia
* known psychiatric disorders including Attention Deficit Disorder
* birth complications needing intensive care
* central nervous system treatment
* important hearing disabilities
* not corrected impaired vision

Ages: 8 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2014-03-18 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Brain area activity in arithmetic processing will be identified by IRMf | up to 60 days after inclusion
  Brain activity is identified by IRMf

SECONDARY OUTCOMES:
Parietal region activity in arithmetic processing will be identified by IRMf | up to 60 days after inclusion
  comparison between group aged to 12to 14 and group aged to 8 to 11

CONTACTS AND LOCATIONS:
Locations (1):
- Médecine nucléaire, Groupement Hospitalier Est, HCL, Bron, France

REFERENCES:
- [Result] Mathieu R, Epinat-Duclos J, Leone J, Fayol M, Thevenot C, Prado J. Hippocampal spatial mechanisms relate to the development of arithmetic symbol processing in children. Dev Cogn Neurosci. 2018 Apr;30:324-332. doi: 10.1016/j.dcn.2017.06.001. Epub 2017 Jun 13. PMID 28648549